CLINICAL TRIAL: NCT05990283
Title: Comparison of Non-grafted Socket Shield Technique With Guided Bone Regeneration in Immediate Implant Placement
Brief Title: Socket Shield Technique and Guided Bone Regeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ezgi Gürbüz, Assistant Professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0044
Record Dates: First submitted 2023-07-29; First posted 2023-08-14 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2019-11

CONDITIONS: Immediate Implant Placement
Keywords: bone regeneration; dental implant; esthetics; grafts; socket shield technique
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Socket shield technique with immediate implant placement (Experimental): For the patients in the shield group, shields were prepared with the Root Membrane Kit. After the palatal part was removed, the buccal fragment was prepared at the crest level, and an internal bevel chamfer was formed on the fragment. Implants were placed 3-4 mm apical to the gingival margin of the adjacent teeth.
  Interventions: Procedure: Socket shield technique
- Guided bone regeneration with immediate implant placement (Experimental): For the patients in the regeneration group, teeth were extracted atraumatically, implants were placed 3-4 mm to the gingival margin, and the space between the implant and buccal bone was filled with anorganic bovine bone graft at the time of implant placement. The graft particles were covered by a pericardium membrane. The membrane was fixed to the bone with titanium pins.
  Interventions: Procedure: Guided bone regeneration

INTERVENTIONS:
Procedure: Socket shield technique — For the patients in the shield group, shields were prepared with the Root Membrane Kit. After the palatal part was removed, the buccal fragment was prepared at the crest level, and an internal bevel chamfer was formed on the fragment. Implants were placed 3-4 mm apical to the gingival margin of the adjacent teeth. Healing caps were placed, and the periphery of the caps was covered with an absorbable gelatin sponge.
  Arms: Socket shield technique with immediate implant placement
Procedure: Guided bone regeneration — For the patients in the regeneration group, teeth were extracted atraumatically, implants were placed 3-4 mm to the gingival margin, and the space between the implant and buccal bone was filled with anorganic bovine bone graft at the time of implant placement. The graft particles were covered by a pericardium membrane. The membrane was fixed to the bone with titanium pins.
  Arms: Guided bone regeneration with immediate implant placement

SUMMARY:
Among the individuals who applied to the Department of Periodontology, Faculty of Dentistry, Health Sciences University between 2019 and 2021, patients with an unrestorable tooth in the maxillary esthetic region and required implant placement were included in this randomized clinical trial. Before implant surgery, patients were randomized into socket shield technique and guided bone regeneration groups. While the buccal gap was untreated in the socket shield group, a xenograft, and membrane were applied in the regeneration group. Peri-implant pocket depth, modified plaque index, modified bleeding index, keratinized mucosa width, and mucosal thickness were recorded at the permanent restoration and the postoperative first year. Horizontal bone level and vertical bone level were assessed with cone beam computed tomography images taken before the surgery and one year after prosthesis insertion. The pink esthetic score was evaluated with intraoral photographs taken before the surgical procedure and first-year follow-up.

DETAILED DESCRIPTION:
This study aimed to compare the non-grafted socket shield technique with simultaneously guided bone regeneration in immediate implant placement in terms of clinical, esthetic, and radiographic parameters. Within the scope, immediate implant placement was applied to randomized groups (socket shield technique and guided bone regeneration). Immediate implant placement was performed following shield preparation in the shield group, and guided bone regeneration was applied in the regeneration group. A temporary non-functional immediate prosthesis was inserted at the same visit. After four months, permanent restorations were applied. Clinical, radiographic, and esthetic parameters were compared between two groups at baseline and first-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the health status of American Society of Anesthesiologists class I or II,
* Nonsmokers,
* Unrestorable single-rooted tooth in the maxillary esthetic region,
* Periodontally healthy, non-mobile teeth,
* Single implant placement,
* Minimum 3-5 mm available vertical bone apical to the apex,
* Intact socket wall after extraction.

Exclusion Criteria:

* Medically compromised patients, especially uncontrolled diabetes,
* Psychiatric problems,
* Pregnancy, lactation, or suspicion of pregnancy,
* A history of radiation therapy to the head and neck region or immunosuppressive therapy,
* Metabolic bone disorder or the presence of drugs known to affect bone metabolism,
* Poor plaque control,
* Vertical root fracture on the buccal surface or a horizontal fracture below the bone level,
* External or internal resorption affecting the buccal part of the root,
* Acute infection in the area intended for implant placement,
* Refusal to attend follow-up appointments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Peri-implant probing depth | Four months after implant restoration and first-year follow-up
  Probing depth measured by Williams periodontal probe
Modified plaque index | Four months after implant restoration and first-year follow-up
  An index evaluated by the Williams periodontal probe indicates a minimum of 0 and a maximum of 3, with higher values indicating a worse outcome
Modified bleeding index | Four months after implant restoration and first-year follow-up
  An index evaluated by the Williams periodontal probe indicates a minimum of 0 and a maximum of 3, with higher values indicating a worse outcome
Keratinized mucosa width | Four months after implant restoration and first-year follow-up
  The distance from the peri-implant mucosa margin to the mucogingival junction
Mucosal thickness | Four months after implant restoration and first-year follow-up
  The thickness measured at 1.5 mm from the margin by the endodontic spreader
Radiographic bone level in the horizontal dimension | Before implant surgery and first year follow-up
  Horizontal bone level measured at cone beam computed tomography images
Radiographic bone level in the vertical dimension | Before implant surgery and first year follow-up
  Vertical bone level measured at cone beam computed tomography images
Pink esthetic score | Before implant surgery and first year follow-up
  A score as assessed by intraoral photographs, showing a minimum of 0 and a maximum of 14, with higher values indicating a better esthetic result

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Ceylan, PhD, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No